CLINICAL TRIAL: NCT00560079
Title: A Double-blind, Randomized, Placebo-controlled 4-week Study on the Efficacy and Safety of the Purinergic Agents Allopurinol and Dipyridamole in Acute Bipolar Mania.
Brief Title: Efficacy of Allopurinol and Dypiridamole in Acute Mania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Espirita de Porto Alegre (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03T-356
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Mania
MeSH Terms: conditions — Mania | interventions — Allopurinol; Dipyridamole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Lithium 900mg/day plus allopurinol 600mg/day
  Interventions: Drug: Allopurinol
- 2 (Active Comparator)
  Interventions: Drug: Dipyridamole
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol — Allopurinol 600mg/day bid for 28 days
  Arms: 1
Drug: Dipyridamole — Dipyridamole 200mg/day bid for 28 days
  Arms: 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
This study aims to evaluate the potential antimanic efficacy, safety and tolorability of the purinergic agents allopurinol and dipyridamole as an add-on treatment to lithium in a sample of 180 drug-free manic patients enrolled in a double-blind, placebo-controlled design.

DETAILED DESCRIPTION:
Men and women ages 18 to 65 years, who were inpatients with a diagnosis of manic episode were recruited at the emergency room of Espirita Hospital of Porto Alegre (HEPA), Brazil (n=180) between September 2004 and 2006. The presence of manic episode was confirmed using SCID-I and the severity of episode was evaluated using the Young Mania Rating Scale (YMRS) and the Clinical Global Impression scale (CGI). Patients were required to present a score>22 on the YMRS at screening to be included. Subjects presenting rapid cycling, mixed episodes and comorbidities with axis I psychiatric disorders were not considered for inclusion. All subjects presented good physical health determined by physical exam, medical history, blood screening and electrocardiogram. Patients were randomly assigned to allopurinol 600 mg/day, dipyridamole 200mg or placebo as add-on medication lithium treatment for a 4-week, double-blind trial. The use of adjunctive antipsychotic agents (typical or second-generation drugs) was not allowed during the double-blind period. Adjunctive diazepam was used when necessary (maximum dose=20mg/day). Raters (psychiatrists) were trained together to establish reliability (YMRS =0.90). This study was approved by the Espirita Hospital Ethics Committee-IRB. Written informed consent was obtained from all patients and/or family member. Possible adverse events were monitored weekly during the follow-up period. Regarding primary outcome measures, we compared the percentage of responders according YMRS score decrease of at least 50% among allopurinol, dipyridamole and placebo groups, using fisher exact test. Also, the percentage of improvement from baseline to endpoint was obtained and compared among groups using analysis of variances (one-way ANOVA) with Duncan post-hoc test. Remission rates (YMRS scores < 12) were also analyzed. P values < 0.05 were considered statistically significant. Besides completers analysis, intention to treat and LOCF were employed to include data from drop-out patients who were evaluated at visit 3. Possible correlations were measured using Pearson test. Fischer exact test and X2 evaluated response and remission rates. Data are presented as mean ± standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* The presence of manic episode was confirmed using SCID-I and the severity of episode was evaluated using the Young Mania Rating Scale (YMRS) and the Clinical Global Impression scale (CGI). Patients were required to present a score>22 on the YMRS at screening to be included.All subjects presented good physical health determined by physical exam, medical history, blood screening and electrocardiogram

Exclusion Criteria:

* Subjects presenting rapid cycling, mixed episodes and comorbidities with axis I psychiatric disorders were not considered for inclusion. .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2003-11; Primary Completion 2005-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
This study aimed to evaluate the potential antimanic efficacy, safety and tolerability | 28 days

SECONDARY OUTCOMES:
Plasma uric acid levels | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Machado-Vieira, MD, MSc, PhD, Principal Investigator — Staff Member
Locations (1):
- Hospital Espirita de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Machado-Vieira R, Soares JC, Lara DR, Luckenbaugh DA, Busnello JV, Marca G, Cunha A, Souza DO, Zarate CA Jr, Kapczinski F. A double-blind, randomized, placebo-controlled 4-week study on the efficacy and safety of the purinergic agents allopurinol and dipyridamole adjunctive to lithium in acute bipolar mania. J Clin Psychiatry. 2008 Aug;69(8):1237-45. doi: 10.4088/jcp.v69n0806. PMID 18681754